CLINICAL TRIAL: NCT00579410
Title: Evaluation of Esophageal and Gastric Acid Levels in Patients Presenting With Upper Gastrointestinal Symptoms Using a Novel PH System
Brief Title: Comparison of Acid Reflux at Two Levels in the Esophagus Using the BRAVO Capsule
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Responsible Party: Prateek Sharma, MD, Department of Veterans Affairs Medical Center
Organization: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Other Study IDs: PS0019
Record Dates: First submitted 2007-12-21; First posted 2007-12-24 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Esophagitis; Inflammation; Gastritis; Abdominal Pain; Heartburn
Keywords: gastric acid; esophageal reflux; peptic ulcer; heartburn
MeSH Terms: conditions — Esophagitis; Inflammation; Gastritis; Abdominal Pain; Heartburn; Gastroesophageal Reflux; Peptic Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: Patients with Barrett's Esophagus
- B: Patients with reflux symptoms but no Barrett's Esophagus
- C: Patients without reflux symptoms and a normal endoscopy

SUMMARY:
The purpose of this research is to study the level of acid exposure above the gastroesophageal junction and the distal esophagus in patients with reflux symptoms using a capsule type acid measurement system. Patients with reflux symptoms are likely to have more acid reflux just above the junction of the stomach and the esophagus that may help to improve the diagnosis of gastroesophageal reflux disease (GERD). This may help better treat the reflux symptoms.

DETAILED DESCRIPTION:
Upper gastrointestinal symptoms and diseases, specifically dyspepsia and acid reflux are common problems faced by the adult U.S. population. These symptoms frequently necessitate an upper gastrointestinal endoscopy, which is performed to rule out anatomic diseases. Moreover, these symptoms can be associated with complications such as erosive esophagitis, Barrett's esophagus, peptic ulcer disease and gastric cancer. The role and the level of acid (pH levels) in patients presenting with these symptoms has been poorly defined in previous studies since they have used catheter based pH systems which provided recordings only for 24 hours, at only a single location in the esophagus or stomach, and has been associated with patient discomfort leading to inconsistent results. This pilot project will attempt to study the level of acid exposure in the distal esophagus and proximal stomach of patients and correlate it with their symptoms.

Many individuals in the Western world are troubled by heartburn, acid regurgitation, abdominal pain (dyspepsia), or bowel habit disturbances; up to one in two subjects in cross sectional population based studies report such symptoms. Gastro-esophageal reflux (GERD) is probably the commonest chronic disease of the population of the Western world. The reported prevalence of symptomatic GERD has ranged, on average, from 15% to 25%. Similarly, dyspepsia is a common condition in the general population; the reported prevalence range in populations is 15-40%. The majority of patients have functional (or non-ulcer) dyspepsia in that they do not have any underlying structural explanation for their symptoms, such as peptic ulcer disease or reflux esophagitis. However, given the significant morbidity and absence from work associated with the condition, the pathogenesis and treatment of patients with dyspepsia still requires further research. Studies are thus needed to determine the long term effects of these symptoms on healthcare costs but in the short run to determine the correlation of symptoms to acid levels and acid exposure.

Upper Gastrointestinal Diseases & pH Recording: Continuous esophageal pH recordings are widely used to study GERD and its treatment (5). Gastric pH recordings are less used clinically, but monitoring of gastric pH has been used for the pharmacological comparison of various anti-secretory agents. Continuous pH recordings in the esophagus and stomach are usually displayed as graphs of pH versus time or as percentage of time with pH above or below a particular value (often 4.0).

Although there is no doubt that gastric acidity is directly involved in GERD pathogenesis, relationships between gastric and esophageal acidity are not clear. Lack of focus on gastric acid may relate to the general belief that gastric acid secretion is usually normal in GERD. Distinct patterns of esophageal acidity in GERD have been previously reported. There is a clear relationship between these descriptors and the present findings of integrated esophageal acidity. Previous pH-based analyses have nicely correlated esophagitis grade with acid exposure, but gastric acidity has been somewhat neglected as the major determinant of esophageal acid exposure in GERD aside from observations that acid inhibition could diminish esophageal acid exposure. Hirschowitz reported basal and pentagastrin-stimulated gastric acid secretion in esophagitis comparable to unspecified medical conditions without esophagitis. Others, however, have reported increased basal, peak, or maximal gastric acid secretion in GERD compared to healthy subjects. In studies of gastro-esophageal reflux, the esophageal pH electrode is traditionally positioned above the proximal limit of the lower esophageal sphincter (LES). This convention was adopted early on to avoid the electrode slipping into the stomach during swallowing when the esophagus shortens by 2-3 cm. As consequence, a conventionally placed electrode will only detect acid refluxing into the distal esophagus if it reaches this point 5 cm above the LES. If acid exposure of the most distal esophagus and proximal stomach is greater than that of the conventional measuring point proximal to the LES, it could have significance clinically. This reflux in the distal esophagus and proximal stomach may explain the high incidence of metaplasia and neoplasia of the most distal esophagus that occurs in the general population.

Previous studies in patients with dyspepsia have revealed either normal levels of pH or mildly elevated levels in the stomach. The correlation between the symptoms and the acid levels has been tested only in a few previous studies. The most distal esophagus and the gastroesophageal junction is exposed to significant amounts of gastric acid, even in subjects without reflux or dyspeptic symptoms. This is of importance for not only understanding the pathophysiology of these diseases but also for treatment with acid suppressive medication. Data are lacking on the benefits of effective acid inhibition with proton pump inhibitors in dyspepsia. In two large, double blind multicenter clinical trials, BOND and OPERA , patients (n=1262) with functional dyspepsia were randomized to four weeks of treatment with omeprazole 20 mg or 10 mg once daily, or placebo. The primary efficacy variable was complete absence of symptoms. The BOND but not the OPERA trial showed a significant benefit of omeprazole over placebo. Pooling the BOND and OPERA trials, complete relief of symptoms was achieved in 38.2% of the 20 mg omeprazole group (p=0.002) and in 36.0% of the 10 mg omeprazole group (p=0.02) compared with 28.2% in the placebo group suggesting that acid suppression may play a role in the treatment of these symptoms. However, before future treatment studies are conducted, correlation of patient symptoms with levels of esophageal and gastric pH levels will be important.

Current practice for measuring esophageal and gastric pH: The current catheter based 24-hr pH system involves placement of a catheter into the esophagus and stomach via the nostril. The tip of the catheter has sensors to measure esophageal and gastric pH. The patient is then sent home (after the catheter is placed, tip coming out of one nostril) and is given a box that measures pH exposure. This is uncomfortable to the patient, leading to change in their daily activities, diet, etc. with resulting data probably not reflective of their "daily habits". Moreover, since the catheter is passed blindly into the esophagus and stomach, the exact location of pH measurement is probably not accurate.

The Bravo pH System: The Bravo pH system (FDA approved) is a novel capsule based and wireless testing system, which allows a capsule, size of a kidney bean, to be attached in the esophagus or the stomach once the endoscopy has been performed. This attachment is helped with the use of a small clip, which then detaches and is passed through the patient in the stool. Preliminary studies using this Bravo pH capsule have shown good tolerability of using this, presence of 48-hour results as well as good correlation with acid suppressive therapy in these patients. To study the level of acid exposure in the stomach and the distal esophagus in patients with upper gastrointestinal diseases and symptoms, specifically in those with dyspepsia and acid reflux using a novel pH system.

Study Design: Patients presenting to the gastroenterology endoscopy unit for upper gastrointestinal symptoms will be invited to participate in the study. The patient's symptoms will be accurately noted using standardized and validated questionnaires. All patients will undergo standard upper endoscopy. The patient demographics including age, gender, ethnicity will be noted. The findings at the time of upper endoscopy such as presence of hiatal hernia, erosive esophagitis, ulcer disease, H. pylori infection, and cancer will be recorded. After the endoscopic procedure is over, two Bravo pH capsules will be placed in the distal esophagus and the proximal stomach after the landmarks have been determined endoscopically. The patients will be provided with a single pH recorder and will be asked to return to the Gastroenterology unit lab, 24-48 hours after placement. Patients will be encouraged to continue with their routine activity including meals. They will fill out a second questionnaire at the end of the study regarding any discomfort that they may have experienced with the Bravo capsule. Data will then be recorded regarding the levels of acid exposure at the sites in the esophagus and stomach, patient demographics and comfort.

Safety Evaluation: Patients who have undergone Bravo in previous studies have reported chest discomfort, chest pain, abdominal pain, and nausea. No major complications have been reported. Thus, there is not a significant risk to the patient undergoing the procedure, except that of the standard endoscopy, for which they have already been scheduled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred for upper endoscopy for any reason including those with acid reflux, dyspepsia, weight loss, Barrett's esophagus,suspected Helicobacter pylori infection.
2. Patients able to provide written informed consent.

Exclusion Criteria:

1. Lack of severe comorbid conditions precluding an upper endoscopy.
2. Patients with history of esophageal or gastric cancer.
3. Patients status post esophageal or gastric resection.
4. Patients with esophageal varices.
5. Patients with severe esophageal strictures.
6. Patients with acute upper gastrointestinal bleeding.
7. Inability to provide informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects in this study were selected from veterans ages 18 and above presenting for an upper endoscopy
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2004-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
This pilot project will attempt to study the level of acid exposure in the distal esophagus and proximal stomach of patients and correlate it with their symptoms. | 24 hour period

SECONDARY OUTCOMES:
To note patient satisfaction and comfort during the pH monitoring process. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Department of Veterans Affairs Medical Center of Kansas City
Locations (1):
- Department of Veterans Affairs Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Background] Talley NJ, Zinsmeister AR, Schleck CD, Melton LJ 3rd. Dyspepsia and dyspepsia subgroups: a population-based study. Gastroenterology. 1992 Apr;102(4 Pt 1):1259-68. PMID 1551533
- [Background] Talley NJ, Phillips SF. Non-ulcer dyspepsia: potential causes and pathophysiology. Ann Intern Med. 1988 Jun;108(6):865-79. doi: 10.7326/0003-4819-108-6-865. PMID 3285748
- [Background] Locke GR 3rd, Talley NJ, Fett SL, Zinsmeister AR, Melton LJ 3rd. Prevalence and clinical spectrum of gastroesophageal reflux: a population-based study in Olmsted County, Minnesota. Gastroenterology. 1997 May;112(5):1448-56. doi: 10.1016/s0016-5085(97)70025-8. PMID 9136821
- [Background] Agreus L. Natural history of dyspepsia. Gut. 2002 May;50 Suppl 4(Suppl 4):iv2-9. doi: 10.1136/gut.50.suppl_4.iv2. PMID 11953337
- [Background] Jamieson JR, Stein HJ, DeMeester TR, Bonavina L, Schwizer W, Hinder RA, Albertucci M. Ambulatory 24-h esophageal pH monitoring: normal values, optimal thresholds, specificity, sensitivity, and reproducibility. Am J Gastroenterol. 1992 Sep;87(9):1102-11. PMID 1519566
- [Background] Robertson D, Aldersley M, Shepherd H, Smith CL. Patterns of acid reflux in complicated oesophagitis. Gut. 1987 Nov;28(11):1484-8. doi: 10.1136/gut.28.11.1484. PMID 3428675
- [Background] Johnston BT, Collins JS, McFarland RJ, Love AH. Are esophageal symptoms reflux-related? A study of different scoring systems in a cohort of patients with heartburn. Am J Gastroenterol. 1994 Apr;89(4):497-502. PMID 8147349
- [Background] Bell NJ, Burget D, Howden CW, Wilkinson J, Hunt RH. Appropriate acid suppression for the management of gastro-oesophageal reflux disease. Digestion. 1992;51 Suppl 1:59-67. doi: 10.1159/000200917. PMID 1397746
- [Background] Hirschowitz BI. A critical analysis, with appropriate controls, of gastric acid and pepsin secretion in clinical esophagitis. Gastroenterology. 1991 Nov;101(5):1149-58. doi: 10.1016/0016-5085(91)90062-p. PMID 1936784
- [Background] Hirschowitz BI. Gastric secretion of acid and pepsin in patients with esophageal stricture and appropriate controls. Dig Dis Sci. 1996 Nov;41(11):2115-22. doi: 10.1007/BF02071389. PMID 8943961
- [Background] Hirschowitz BI. Gastric acid and pepsin secretion in patients with Barrett's esophagus and appropriate controls. Dig Dis Sci. 1996 Jul;41(7):1384-91. doi: 10.1007/BF02088563. PMID 8689915
- [Background] Collen MJ, Lewis JH, Benjamin SB. Gastric acid hypersecretion in refractory gastroesophageal reflux disease. Gastroenterology. 1990 Mar;98(3):654-61. doi: 10.1016/0016-5085(90)90285-9. PMID 2298369
- [Background] Gillen P, Keeling P, Byrne PJ, Hennessy TP. Barrett's oesophagus: pH profile. Br J Surg. 1987 Sep;74(9):774-6. doi: 10.1002/bjs.1800740906. PMID 3664238
- [Background] Gardner JD, Rodriguez-Stanley S, Robinson M. Integrated acidity and the pathophysiology of gastroesophageal reflux disease. Am J Gastroenterol. 2001 May;96(5):1363-70. doi: 10.1111/j.1572-0241.2001.03790.x. PMID 11374669
- [Background] Fletcher J, Wirz A, Henry E, McColl KE. Studies of acid exposure immediately above the gastro-oesophageal squamocolumnar junction: evidence of short segment reflux. Gut. 2004 Feb;53(2):168-73. doi: 10.1136/gut.2003.022160. PMID 14724145
- [Background] Samsom M, Verhagen MA, vanBerge Henegouwen GP, Smout AJ. Abnormal clearance of exogenous acid and increased acid sensitivity of the proximal duodenum in dyspeptic patients. Gastroenterology. 1999 Mar;116(3):515-20. doi: 10.1016/s0016-5085(99)70171-x. PMID 10029608
- [Background] George AA, Tsuchiyose M, Dooley CP. Sensitivity of the gastric mucosa to acid and duodenal contents in patients with nonulcer dyspepsia. Gastroenterology. 1991 Jul;101(1):3-6. doi: 10.1016/0016-5085(91)90453-r. PMID 2044924
- [Background] Collen MJ, Loebenberg MJ. Basal gastric acid secretion in nonulcer dyspepsia with or without duodenitis. Dig Dis Sci. 1989 Feb;34(2):246-50. doi: 10.1007/BF01536059. PMID 2914546
- [Background] Talley NJ, Lauritsen K. The potential role of acid suppression in functional dyspepsia: the BOND, OPERA, PILOT, and ENCORE studies. Gut. 2002 May;50 Suppl 4(Suppl 4):iv36-41. doi: 10.1136/gut.50.suppl_4.iv36. PMID 11953346
- [Background] Veldhuyzen van Zanten SJ, Cleary C, Talley NJ, Peterson TC, Nyren O, Bradley LA, Verlinden M, Tytgat GN. Drug treatment of functional dyspepsia: a systematic analysis of trial methodology with recommendations for design of future trials. Am J Gastroenterol. 1996 Apr;91(4):660-73. PMID 8677926
- [Background] Talley NJ. Review article: functional dyspepsia--should treatment be targeted on disturbed physiology? Aliment Pharmacol Ther. 1995 Apr;9(2):107-15. doi: 10.1111/j.1365-2036.1995.tb00359.x. PMID 7605850
- [Background] 23. Carlsson R, Bolling E, Jerndal , et al. Factors predicting response to omeprazole treatment in patients with functional dyspepsia. Gastroenterology 1996;110:A76.